CLINICAL TRIAL: NCT07156305
Title: College Student Alcohol Behaviors and Strategies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Anna Michelle Petrey, Clinical Psychology Doctoral Student, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-2025-254
Record Dates: First submitted 2025-08-26; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use
Keywords: Protective behavioral strategy; PBS; Protective behavioral strategies; Alcohol use; Alcohol consequences
MeSH Terms: conditions — Alcohol Drinking | interventions — Organizational Objectives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants complete measures at baseline and follow-up, and receive psychoeducation on PBS.
- PBS-only (Active Comparator): Participants complete measures at baseline and follow-up, receive psychoeducation about PBS, select three PBS strategies, and select a reminder strategy.
  Interventions: Behavioral: Protective Behavioral Strategies
- PBS+Goals (Experimental): Participants complete measures at baseline and follow-up, receive psychoeducation about PBS and goal-setting, select three PBS strategies, select two goals related to each PBS strategy chosen, and select a reminder strategy.
  Interventions: Behavioral: Goal-Setting

INTERVENTIONS:
Behavioral: Protective Behavioral Strategies — Participants receive psychoeducation about protective behavioral strategies and are asked to choose three strategies that they do not already engage in regularly but would be willing to start using more.
  Arms: PBS-only
Behavioral: Goal-Setting — Participants receive psychoeducation about protective behavioral strategies and goal-setting. They are asked to choose three strategies that they do not already engage in regularly and identify two goals related to each strategy.
  Arms: PBS+Goals

SUMMARY:
The primary goal of this clinical trial is to examine whether the use of personalized goal setting related to protective behavioral strategies (PBS)-behavioral techniques enacted before, during, or after alcohol consumption to reduce risk and minimize harm-increases the use of personally selected PBS implementation. A secondary goal of this trial is to examine whether increasing the frequency of PBS use will lead to decreases in alcohol consumption, fewer alcohol-related negative consequences, and increased alcohol-related positive consequences. Researchers will compare a control condition, a PBS-only condition, and a PBS+Goals condition to address the aims of the study. Participants in all conditions will complete measures about current PBS use, alcohol use and consequences, and likelihood and confidence to change current alcohol and strategy use. All participants will receive brief psychoeducation on PBS. Participants in the PBS-only and PBS+Goals condition will select three PBS to use over the following two weeks, and select a strategy for remembering the PBS they chose. Participants in the PBS+Goals condition will receive psychoeducation about goal setting and identify two goals related to each PBS strategy they selected. Participants in all conditions will complete a follow-up after two weeks containing measures about PBS use, alcohol use and consequences, and likelihood and confidence to change alcohol and strategy use. Participants in the PBS-only and PBS+Goals condition will complete a measure to indicate whether they used the reminder strategy they selected at the two-week follow-up. Participants in the PBS+Goals condition will complete a measure indicating whether they believe they achieved their goals at the two-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Must report being between the ages of 18-25
* Must report engaging in alcohol use at least one time per week over the past two weeks, on average

Exclusion Criteria:

* Reports currently receiving or having received treatment for their alcohol or other substance use during the past two months
* Age below 18 or above 25 years
* Does not report having engaged in alcohol use at least one time per week over the past two weeks, on average

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Protective Behavioral Strategy Use | Baseline and two-week follow-up.
  Participants will be asked at baseline and follow-up to indicate the frequency they use the various PBS included in the Protective Behavioral Strategies Scale - 20 (PBSS-20) across the past two weeks. Change will be examined across groups as the mean change in past-two-week frequency of PBS use at follow-up relative to baseline.
Alcohol Use | Baseline and two-week follow-up
  Participants will be asked to complete the Timeline Follow-Back (TLFB), a measure of past-two-week alcohol use, at baseline and follow-up. Change will be examined across groups as mean change in past-two-week alcohol use at at follow-up relative to baseline.
Negative Alcohol-Related Consequences | Baseline and two-week follow-up
  Participants will be asked to report on the total number of negative alcohol-related consequences they have experienced in the past two weeks using the Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ). Change will be examined across group as the mean change in number of negative alcohol-related consequences experienced across the past two weeks at follow-up relative to baseline.
Positive Alcohol-Related Consequences | Baseline and two-week follow-up
  Participants will be asked to report on the number of positive alcohol-related consequences they have experienced across the past two weeks at baseline and follow-up using the Positive Drinking Consequences Questionnaire (PDCQ). Change across groups will be examined as the mean change in number of positive alcohol-related consequences at follow-up relative to baseline.

SECONDARY OUTCOMES:
Likelihood to Change | Baseline and two-week follow-up
  Participants will report on the likelihood of them changing their alcohol and PBS use on a scale of 1 (not likely) to 10 (very likely) on a two-item custom measure. Items include: 1. "Please rate how likely you are to make changes to your drinking behaviors, so you drink less or drink in a safer way. Please base the following answer based on how you are feeling RIGHT NOW." and 2. "Please circle how likely you are to try out new strategies to help you drink less or drink more safely. Please base the following answer based on how you are feeling RIGHT NOW." Change will be examined across groups as mean change in likelihood of changing at follow-up relative to baseline.
Confidence in Changing | Baseline and two-week-follow-up
  Participants will report how confident they are in changing their alcohol and PBS use on a scale of 1 (not confident) to 10 (very confident) on a two-item custom measure. Items include: 1. "Please circle how confident you are in your ability to change your drinking, so you drink less or drink in a safer way. Please base the following answer based on how you are feeling RIGHT NOW." and 2. "Please circle how confident you are that you could use new strategies to help you drink less or drink more safely. Please base the following answer based on how you are feeling RIGHT NOW." Change will be examined across groups as mean change in confidence of changing at follow-up relative to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No